CLINICAL TRIAL: NCT04989413
Title: Randomized, Double Blind Clinical Trial to Study the Effect of Cannabidiol (CBD) 133mg + Cannabigerol (CBG) 66mg + Tetrahydrocannabinol (THC) 4mg a Day As Adjunctive Therapy in the Treatment of Chronic Migraine - CAMTREA TRIAL
Brief Title: Cannabidiol 133mg + Cannabigerol 66mg + Tetrahydrocannabinol 4mg Vs Placebo As Adjuvant Treatment in Chronic Migraine -
Acronym: CAMTREA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: an interim analysis to rule out futility was positive, we completed active patients and stopped recruitment with 75 patients enrolled
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Industria Farmacêutica Health Meds (Unknown)
Responsible Party: Principal Investigator, Alexandre Kaup, Principal Investigator, MD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIAE CAMTREA Protocol
Record Dates: First submitted 2021-05-24; First posted 2021-08-04 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Chronic Migraine, Headache; Overuse Headache Medication
MeSH Terms: conditions — Headache; Headache Disorders, Secondary | interventions — Cannabidiol; cannabigerol; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol + Cannabigerol + Tetrahydrocannabinol 133/66/4mg (Active Comparator): Cannabidiol + Cannabigerol + Tetrahydrocannabinol in the maximum dosage of 133/66/4mg, divided in 2 doses of 66.5/33/2mg a day for 12 weeks. Each drop contain CBD/CBG/THC 1.66/0.8/0.05 mg, and medication will be titrated up as follow: day 1 to day 3 - 10 drops twice a day day 4 to day 6 - 20 drrops twice a day day 7 to day 9 - 30 drops twice a day from day 10 to the end of the study 40 drops twice a day
  Interventions: Drug: Cannabidiol + Cannabigerol + Tetrahydrocannabinol 133/66/4mg
- Placebo (Placebo Comparator): Placebo capsules will be titrated up as follow:
  day 1 to day 3 - 10 drops twice a day day 4 to day 6 - 20 drops twice a day day 7 to day 9 - 30 drops twice a day from day 10 to the end of the study 40 drops twice a day
  Interventions: Drug: Placebo oral drops

INTERVENTIONS:
Drug: Placebo oral drops — use of placebo for 12 weeks
  Arms: Placebo
Drug: Cannabidiol + Cannabigerol + Tetrahydrocannabinol 133/66/4mg — use of cannabidiol + canabigerol + thc for 12 weeks
  Arms: Cannabidiol + Cannabigerol + Tetrahydrocannabinol 133/66/4mg

SUMMARY:
To evaluate the effect of the cannabidiol (CBD) + cannabigerol (CBG) + tetrahydrocannabinol (THC) up to 133/66/4mg daily versus placebo as adjuvant treatment in chronic migraine (CM) patients under preventive treatment at a stable dose for at least 3 months who present at least 5 headaches day a month. CM patients of both sexes, between 25 and 65 years old, who have not had CBD and/or THC as a migraine treatment. Patients may be having migraine preventive treatment such as propranolol, atenolol, topiramate, valproic acid/sodium valproate, levetiracetam, gabapentin, lamotrigine, pre-gabaline, flunarizine, amitriptyline, nortriptyline, clomipramine, candesartan, galcanezumab, erenumab, fremanezumab, botulinum toxin type A. Acute treatment will follow patients doctor's prescription. Exclusion criteria: active liver disease or elevated liver transaminases> 3 times than the normal values, pregnancy, fertile age women without contraceptive treatment or who intend to get pregnant, patients without migraine preventive treatment or that changed the preventive treatment less than 3 months from the study start, substance abuse or addiction, use of medical cannabis or products with CBD or THC in the last 30 days or during study period, history of allergy or adverse reactions with the use of CBD or related products, substance users of liver enzymes inducers such as rifampicin, ketoconazole, theophylline, carbamazepine, phenytoin, phenobarbital and St. John's wort, clobazam, macrolides, verapamil, fluoxetine, amiodarone and tacrolimus. Patients on vitamin K anticoagulant medicines, as warfarin.

Randomization using a computacional system will stratify participants in each group by gender (F/M), age (25-34/35-44/45-54/55-65yo), headache days presented in the baseline month (5-10/11-15/16-20/21-25/26-30), overuse medication (yes or no). After randomization patients will be divided into two groups of 55 participants, who will receive CBD + CBG + THC up to a maximum daily dose of 133/66/4 mg or placebo for 12 weeks (V0 screening, V1 allocation, V4 final visit).

The main outcome is the reduction in frequency of headache days per 4 weeks between V1 and V4 compared to placebo. Secondary outcomes will be a reduction in duration and intensity of migraine attacks, amount of painkillers used and percentage of patients with a reduction greater than 50% on migraine days, 50% reduction in the other variables as MIDAS scores, HIT-6 scores, Beck's Anxiety and Depression Scales, Epworth Sleepiness Scales, and the scores at The Severity of Dependence Scale used as an indicator of overuse medication in this sample.

Clinical data will be registered on a personalized headache diary developed to this study using MyCap, from RedCap System, as an APP for daily entries using smartphones, androids or IOS system.

The clinical and laboratory data obtained in this study will comply with the objectives elaborated in the evaluation of the primary and secondary endpoints, the proposal of which is to publish the data regardless of the results obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, 25 to 65 years old, with chronic migraine according to IHS Classification System, 3rd edition
* Undergoing preventive treatment in a stable dose of the preventive medication for at least 2 months, who have not used cannabidiol to treat migraine.
* At least 5 days of migraine/migraine like attacks in the baseline period (4 weeks)
* As preventive drugs propranolol, atenolol, topiramate, valproic acid/sodium valproate, levetiracetam, gabapentin, lamotrigine, pre-gabaline, flunarizine, amitriptyline, nortriptyline, clomipramine, candesartan, galcanezumab, erenumab, fremanezumab, botulinum toxin type A will be allowed. Patients whose preventive treatment for migraine is Botulinum Toxin Type A may participate in the study as long as the toxin application interval used is 4 months (duration of medication or placebo use) and who have already received treatment with toxin at least 2 times.
* If acute treatment is necessary, patients may use the medications as previously advised by the physician accompanying them, and may use common, combined painkillers, anti-inflammatory drugs, triptans, triptans combined with anti-inflammatory drugs, opioid analgesics.

Exclusion Criteria:

* Patients with active liver disease
* pregnancy and/or women who intend to become pregnant or who do not make adequate use of contraceptive therapy/methods
* breastfeeding women
* use of cannabis during the study, whether with therapeutic or recreational intentions
* patients who are without preventive treatment or who have undergone a dose change in preventive migraine treatment less than two months before V1 .
* Patients whose exclusive treatment for chronic migraine is Botulinum Toxin Type A at intervals of less than 4 months.
* History of substance abuse or addiction, use of medical cannabis or products with CBD, CBG or THC in the last 30 days, history of allergy to CBD or related products
* elevated transaminases > 3x the normal value
* substance abusers
* patients using substances that are potent enzyme inducers, such as rifampicin, ketoconazole, theophylline, carbamazepine, phenytoin, phenobarbital and St. John's wort, clobazam, macrolides, verapamil, fluoxetine, amiodarone and tacrolimus.
* Patients using anticoagulant, like vitamin K anticoagulant medicines, as warfarin.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Migraine days | 16 weeks
  The primary outcome will be the reduction in migraine days observed between the baseline period (4 weeks before randomization) and the final visit 12 weeks of intervention (CBD+CBG+THC or placebo)

SECONDARY OUTCOMES:
Headache days | 12 weeks
  The primary outcome will be the reduction in headache days observed between the baseline period (4 weeks before randomization) and the final visit 12 weeks of intervention (CBD+CBG+THC or placebo)
migraine duration | 12 weeks
  the attack duration in hours observed before and after the intervention (CBD+CBG+THC or placebo)
migraine intensity | 12 weeks
  the migraine attack intensity measured in a 3 point scale (1- mild; 2 - moderate; 3 - severe) before and after the intervention (CBD+CBG+THC or placebo)
pain medicine intake | 12 weeks
  the amount of pain medicine intake as needed before and after the intervention (CBD+CBG+THC or placebo)
number of patients with migraine reduction greater than 50% | 12 weeks
  the number of patients with migraine reduction greater than 50% before and after the intervention (CBD+CBG+THC or placebo)
number of patients with headache reduction greater than 50% | 12 weeks
  the number of patients with migraine reduction greater than 50% before and after the intervention (CBD+CBG+THC or placebo)
Change in MIDAS score | 12 weeks
  the observed change in MIDAS score, before and after the intervention (CBD+CBG+THC or placebo)
Change in HIT-6 score | 12 weeks
  the observed reduction in HIT-6 score, before and after the intervention (CBD+CBG+THC or placebo)
Change in Beck's Anxiety Inventory scores | 12 weeks
  the observed change in BAI score, before and after the intervention (CBD+CBG+THC or placebo)
Change in Beck's Depression Inventory scores | 12 weeks
  the observed change in BDI score, before and after the intervention (CBD+CBG+THC or placebo)
Change in Severity of Dependence Scale scores | 12 weeks
  the observed change in SDS score, before and after the intervention (CBD+CBG+THC or placebo)
Change in Epworth Sleepiness Scale scores | 12 weeks
  the observed change in Epworth score, before and after the intervention (CBD+CBG+THC or placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre O Kaup, MD, PhD, Principal Investigator — Clinical Research Hospital Israelita Albert Einstein, Neurologist
Locations (1):
- Centro de Pesquisa Clinica Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No